CLINICAL TRIAL: NCT00690677
Title: Phase II Trial of LBH589 in Refractory Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589BUS19T; CRC GOLP CNOV 0823
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Cancer
Keywords: LBH589; Metastatic Colorectal Cancer; Refractory Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: LBH589 — LBH589 will be administered orally at a dose of 30mg (1 - 20mg capsule and 2 - 5g capsules) on Monday, Wednesday and Friday of each week (three times a week). Patients may continue treatment with oral LBH589 until they experience unacceptable toxicity that precludes further treatment, disease progression, and/or at the discretion of the investigator.
  The LBH589 capsules should be swallowed by mouth with a glass of water in the morning. The recommended way to take LBH589 is after not eating for at least 2 hours. You should also not eat for another 2 hours after taking your LBH589 capsules. The daily dose of LBH589 should be taken at approximately the same time each day. You should avoid eating grapefruit, seville oranges, or drinking grapefruit or seville orange juice during the study.

SUMMARY:
The purpose of this study is to determine the effects of the study drug, LBH589, on patients with metastatic colorectal cancer that has continued to grow despite previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years old
* Patients with measurable metastatic colorectal cancer
* Refractory to at least 2 standard chemotherapy/biologic regimens to include 5FU, oxaliplatin, irinotecan, bevacizumab, cetuximab or combinations thereof
* ECOG Performance Status of ≤ 2
* Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Laboratory values as follows:

  * Neutrophil count of >1500/mm3
  * Platelet count of > 100,000/mm3L
  * Hemoglobin ≥ 9 g/dL
  * AST/SGOT and ALT/SGPT ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement
  * Serum bilirubin ≤ 1.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 ml/min
  * Total serum calcium (corrected for serum albumin) or ionized calcium ≥ LLN
  * Serum potassium ≥ LLN
  * Serum sodium ≥ LLN
  * Serum albumin ≥ LLN or 3g/dl
  * Patients with any elevated Alkaline Phosphatase due to bone metastasis can be enrolled
* Baseline MUGA or ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal
* TSH and free T4 within normal limits (patients may be on thyroid hormone replacement)
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of study treatment. and must be willing to use two methods of contraception one of them being a barrier method during the study and for 3 months after last study drug administration
* Radiographically bi-dimensionally measurable disease that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation
* Life expectancy must be greater than 12 weeks

Exclusion Criteria:

* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
* Impaired cardiac function including any one of the following:

  * Screening ECG with a QTc > 450 msec confirmed by central laboratory prior to enrollment to the study
  * Patients with congenital long QT syndrome
  * History of sustained ventricular tachycardia
  * Any history of ventricular fibrillation or torsades de pointes
  * Bradycardia defined as heart rate < 50 beats per minute. Patients with a pacemaker and heart rate ≥ 50 beats per minute are eligible.
  * Patients with a myocardial infarction or unstable angina within 6 months of study entry
  * Congestive heart failure (NY Heart Association class III or IV)
  * Right bundle branch block and left anterior hemiblock (bifasicular block)
* Uncontrolled hypertension
* Concomitant use of drugs with a risk of causing torsades de pointes
* Concomitant use of CYP3A4 inhibitors
* Patients with unresolved diarrhea > CTCAE grade 1
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
* Other concurrent severe and/or uncontrolled medical conditions
* Patients who have received chemotherapy, any investigational drug or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
* Concomitant use of any anti-cancer therapy or radiation therapy
* Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of oral LBH589
* Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom
* Patients with a history of another primary malignancy within 5 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
* Patients with known positivity for human immunodeficiency virus (HIV) ) or hepatitis C; baseline testing for HIV and hepatitis C is not required
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of LBH589 on overall survival (OS) in patients with colorectal cancer | 18 months

SECONDARY OUTCOMES:
Time to tumor progression and response rates | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gold, MD, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States